CLINICAL TRIAL: NCT06710080
Title: Targeting Vascular INflammation in Patients with Community-Acquired Pneumonia (TIN_CAP): a Multi-centre, Prospective, Randomized Control Trial
Brief Title: Targeting Vascular INflammation in Patients with Community-Acquired Pneumonia
Acronym: TIN-CAP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-10

CONDITIONS: Inflammation; Community Acquired Pneumonia (CAP); Inflammation Plaque, Atherosclerotic
Keywords: Community-Acquired Infection; Plaque, atherosclerotic; Inflammation; Eicosapentaenoic Acid
MeSH Terms: conditions — Inflammation; Community-Acquired Pneumonia; Community-Acquired Infections; Plaque, Atherosclerotic | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Participants randomized to this arm will receive Vascepa for 6 months.
  Interventions: Drug: Icosapent Ethyl 1000 MG Oral Capsule [Vascepa]
- Placebo (Placebo Comparator): Participants randomized to this arm will receive placebo for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Icosapent Ethyl 1000 MG Oral Capsule [Vascepa] — Participants randomized to the treatment arm will receive Vascepa 1000mg twice a day for 6 months.
  Arms: Treatment
Drug: Placebo — Placebo twice daily
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if icosapent ethyl (Vascepa) works to lessen the amount of inflammation in adults diagnosed with Community-Acquired Pneumonia (CAP). The main question it aims to answer is:

What is the effect of taking Vascepa on inflammation in the arteries in patients with CAP? Researchers will compare the drug Vascepa to a placebo (a look-alike submstance that contains no drug) to see if Vascepa works to reduce inflammation in patients with CAP.

Participants wil:

* take Vacscepa or a placebo twice a day for 6 months
* Visit the clinic 3 times (baseline, 30 days, and 6 months) for checkups and tests

DETAILED DESCRIPTION:
TIN CAP is a multi centre, prospective, randomized, double-blind, placebo-controlled clinical trial to evaluate the use of icosapent ethyl (Vascepa) on vascular inflammation in patients with CAP using FDG-PET/CT imaging and measurement of circulating biomarkers. The current proposal uses a randomized design to:

1. measure the effect of icosapent ethyl vs. placebo on reducing arterial inflammation over a 6-month treatment period, with primary analysis at 6-months;
2. the correlation between imaging and blood biomarkers over time relative to the drug response.

ELIGIBILITY:
Inclusion Criteria:

Patients who have:

1. Hospitalization with CAP (defined as pulmonary infiltration using chest imaging, in addition to other clinical symptoms including fever, cough, and sputum)
2. age > 18 years;
3. given informed consent.

Exclusion Criteria:

Patients who have:

1. history of cancer within the last 3 years (other than a successfully treated cutaneous squamous cell or basal cell carcinoma or localized carcinoma in situ of the cervix).
2. active inflammatory conditions (e.g. rheumatoid arthritis, chronic inflammatory bowel disease, SLE, systemic anti-inflammatory therapy (e.g. prednisone, methotrexate));
3. pregnancy (all women of child bearing potential will have a negative BHCG test;
4. breastfeeding;
5. Women of childbearing potential who refuse to use two forms of contraception (this includes at least one form of highly effective and one effective method of contraception) throughout the study OR men capable of fathering a child who refuse to use contraception.
6. Allergies to icosapent ethyl
7. allergies to fish or shellfish
8. glomerular filtration rate (GFR) <50 ml/min/1.72m2 (excluded from CTA portion)
9. unable to give informed consent;

Exclusion for CTA portion of the protocol:

Patients with dye allergy will not undergo CTA but will have PET/CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The change over 6 months in the FDG uptake TBR as a marker of arterial plaque inflammation between the icosapent ethyl and placebo groups | 6 months

SECONDARY OUTCOMES:
The change in inflammation, measured on FDG PET, in the pulmonary tissue. | 6 months
  The change in background-corrected measure of total metabolic activity (total pulmonary glycolytic activity) will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided